CLINICAL TRIAL: NCT04314505
Title: Opioid-Sparing Protocol Using for Postoperative Pain Management Comparing With Opioid-based Patient Control Analgesia After Simultaneous Bilateral Total Knee Arthroplasty: a Randomized Controlled Trial
Brief Title: Opioid-Sparing Protocol Comparing With Opioid-based Protocol After Bilateral Total Knee Arthroplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-02-008C
Record Dates: First submitted 2020-03-12; First posted 2020-03-19 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Knee Replacement; Postoperative Pain; Opioid Use
Keywords: Bilateral Total Knee Arthroplasty; Opioid Use; Opioid Sparing; Postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Opioid Sparing Protocol (Experimental): Preemptive(before incision): Parecoxib sodium 40 mg Postoperative: Parecoxib sodium 40 mg was given intravenously every 12 hours for 4 more doses.
  Interventions: Drug: Opioid-Sparing Protocol
- Opioid Based Patient Controlled Analgesia (Active Comparator): Preemptive(before incision) and Postoperative: the initial setting was 0.01mg/kg*hour, patient-controlled dose 2 mg, lock-out 5 minutes and limited 40mg in each 4 hours; adjusted by the PCA staff
  Interventions: Drug: Opioid-Based Patient Controlled Analgesia

INTERVENTIONS:
Drug: Opioid-Sparing Protocol — After a general anesthesia procedure was performed, an experienced anesthesiologist performed ultrasound guided adductor canal block procedures on both knees. In the opioid-sparing group, a dose of Parecoxib sodium 40 mg was administrated through intravenous route before the incision. After the surgery, Parecoxib sodium 40 mg was given intravenously every 12 hours for 4 more doses. Before the wound closure, the periarticular injection (each side 10 ml of 0.25% Bupivacaine) was done. The total dosage would be recorded in the device. All patients received oral paracetamol 500mg, 4 times a day and oral celecoxib 200mg, 2 times a day after surgery.
  Other Names: OSP Protocol
  Arms: Opioid Sparing Protocol
Drug: Opioid-Based Patient Controlled Analgesia — After a general anesthesia procedure was performed, an experienced anesthesiologist performed ultrasound guided adductor canal block procedures on both knees. The patient was informed that the intravenous bolus of rescue morphine (4mg) was available every 4 hours if the pain was intolerable. In the PCA group, the device was applied before incision and the initial setting was 0.01mg/kg*hour, patient-controlled dose 2 mg, lock-out 5 minutes and limited 40mg in each 4 hours. After the surgery, the staff of PCA group would visit the patients and adjusted the dosage. The PCA was removed after 72 hours from the surgery. Before the wound closure, the periarticular injection (each side 10 ml of 0.25% Bupivacaine) was done. The total dosage would be recorded in the device. All patients received oral paracetamol 500mg, 4 times a day and oral celecoxib 200mg, 2 times a day after surgery.
  Other Names: PCA Protocol
  Arms: Opioid Based Patient Controlled Analgesia

SUMMARY:
The concern for the opioid use in the total knee arthroplasty continues to rise in recent decades. Historically, the total knee arthroplasty consumed high doses opioids in the postoperative periods. Compared to the Opioid-Based patient controlled analgesia(PCA), the opioid-sparing protocol may have benefits to decrease the concerns of the opioid use and opioid-related complication and provides the equivalent efficacy for pain control. The purpose of this trial in to provide a novel opioid-sparing protocol (OSP) to evaluate the efficacy for pain control and reducing the immediate postoperative opioid consumption.

ELIGIBILITY:
Inclusion Criteria:

* patient with bilateral advanced knee osteoarthritis undergoing simultaneous bilateral total knee arthroplasty surgery
* willing to participate in this study and randomly allocated to either opioid-sparing protocol or PCA protocol.

Exclusion Criteria:

* patient who refused to participate or with contraindication or hypersensitivity to any of the study drugs
* chronic pain disorder (exceeding 50 mg oral morphine equivalence per day at time of recruitment)
* substance abuse (e.g. alcoholism)
* severe renal impairment.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2020-03-20 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2020-08-20 (Estimated)

PRIMARY OUTCOMES:
Pain scores using numerical rating scale (VAS, 0 to 10) at rest | Post-operative 6 hours after surgery
  Post-operative 6 hours
Pain scores using numerical rating scale (VAS, 0 to 10) at rest | Post-operative 12 hours after surgery
  Post-operative 12 hours
Pain scores using numerical rating scale (VAS, 0 to 10) at rest | Post-operative 24 hours after surgery
  Post-operative 24 hours
Pain scores using numerical rating scale (VAS, 0 to 10) at rest | Post-operative 48 hours after surgery
  Post-operative 48 hours
Pain scores using numerical rating scale (VAS, 0 to 10) at rest | Post-operative 72 hours after surgery
  Post-operative 72 hours
Pain scores using numerical rating scale (VAS, 0 to 10) at motion | Post-operative 24 hours after surgery
  Post-operative 24 hours
Pain scores using numerical rating scale (VAS, 0 to 10) at motion | Post-operative 48 hour hours after surgery
  Post-operative 48 hours
Pain scores using numerical rating scale (VAS, 0 to 10) at motion | Post-operative 72 hour hours after surgery
  Post-operative 72 hours

SECONDARY OUTCOMES:
maximum angle of continuous passive motion (CPM) as tolerated (Degrees) | 0-72 hours after surgery
  recorded at post-operative 24 hours, 48 hours and 72 hours
Cumulative morphine consumption(mg) | 0-72 hours after surgery
  recorded at post-operative 24 hours, 48 hours and 72 hours
drug-related (opioid) adverse events | 0-72 hours after surgery
  nausea/vomiting, dizziness, urinary retention, pruritus, dry mouth, constipation, dyspepsia, GI bleeding, pitting edema over lower extremities, cardiovascular event, respiratory depression, delirium or coma
Satisfaction scale (0-100 points) | postoperative 2 weeks after surgery
  satisfaction with regard to the efficacy and safety of the pain management protocol.
Length of hospital stay (LOS) (Days) | After surgery until discharge (about 3-5 days after surgery)
  Time from admission to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Shang-Wen Tsai, M.D., Study Director — Department of Orthopaedic and Traumatology, Taipei Veterans General Hospital
Locations (1):
- Dep. of Orthopedics and Traumatology, Taipei Veterans General Hospital, Taipei City, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No